CLINICAL TRIAL: NCT03210259
Title: VOLTAIRE-X: Pharmacokinetics, Safety, Immunogenicity and Efficacy of BI 695501 Versus Humira® in Patients With Moderate to Severe Chronic Plaque Psoriasis: a Randomized, Double-blind, Parallel-arm, Multiple-dose, Active Comparator Trial
Brief Title: The VOLTAIRE-X Trial Looks at the Effect of Switching Between Humira® and BI 695501 in Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1297-0009; 2016-002254-20 (EudraCT Number)
Record Dates: First submitted 2017-07-05; First posted 2017-07-06 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab; BI 695501

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 695501 (Experimental)
  Interventions: Drug: BI 695501
- Humira® (Active Comparator)
  Interventions: Drug: Humira®

INTERVENTIONS:
Drug: Humira® — Duration - 58 weeks
  Arms: Humira®
Drug: BI 695501 — Duration - 58 weeks
  Other Names: CYLTEZO
  Arms: BI 695501

SUMMARY:
The primary objective of the trial is to assess the PK similarity between patients receiving Humira® continuously vs those who alternate between BI 695501 and Humira®, in patients with moderate-to-severe chronic plaque psoriasis.

The secondary objectives of this trial are to descriptively compare the safety, immunogenicity and efficacy profiles between patients receiving Humira® continuously vs those who alternate between BI 695501 and Humira®.

ELIGIBILITY:
Inclusion criteria

* Males and females aged ≥ 18 to < 80 years at screening who have a diagnosis of moderate-to-severe chronic plaque psoriasis (with or without psoriatic arthritis) for at least 6 months before the first administration of trial drug (a self-reported diagnosis confirmed by the Investigator is acceptable), and which has been stable per Investigator opinion for the last 2 months with no changes in morphology or significant flares at both screening and baseline:

  * involved body surface area (BSA) ≥ 10% and
  * PASI score ≥ 12 and
  * sPGA score of ≥ 3.
* Participants of reproductive potential (childbearing potential1) must be willing and able to use highly effective methods of birth control per International Council for Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly during the trial and for 6 months following completion or discontinuation from the trial medication. A list of contraception methods meeting these criteria is provided in patient information.
* Signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to admission to the trial.
* Patients who are candidates for systemic therapy or phototherapy according to Investigator judgement.

Exclusion criteria

* Active ongoing inflammatory diseases other than psoriasis that might confound trial evaluations according to Investigator's judgment.
* Prior exposure to any biologic therapies for any auto-immune diseases (eg: RA, Psoriasis, Crohns Disease, etc).
* Patients with a significant disease other than psoriasis and/or a significant uncontrolled disease (such as, but not limited to, nervous system, renal, hepatic, endocrine, hematological, autoimmune or gastrointestinal disorders). A significant disease is defined as a disease which, in the opinion of the Investigator, may (i) put the patient at risk because of participation in the trial, or (ii) influence the results of the trial, or (iii) cause concern regarding the patient's ability to participate in the trial.
* Major surgery (major according to the Investigator's assessment) performed within 12 weeks before enrollment or planned within 6 months after screening, e.g., total hip replacement.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated (in the opinion of the Investigator) basal cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Currently enrolled in another investigational device or drug trial, or less than 30 days (or less than 5 half-lives, whichever is longer) since ending another investigational device or drug trial(s), or receiving other investigational treatment(s).
* Chronic alcohol or drug abuse or any condition that, in the Investigator's opinion, makes the patient an unreliable trial subject or unlikely to complete the trial.
* Women who are pregnant, nursing, or who plan to become pregnant during the course of this trial or within the period at least 6 months following completion or discontinuation from the trial medication.
* Forms of psoriasis (e.g., pustular, erythrodermic and guttate) other than chronic plaque psoriasis. Drug-induced psoriasis (i.e., new onset or current exacerbation from e.g., beta blockers or lithium).
* Primary or secondary immunodeficiency (history of, or currently active), including known history of HIV infection or a positive HIV test at screening (per the Investigator discretion and where mandated by local authorities).
* Known chronic or relevant acute TB; IGRA TB test or PPD skin test will be performed according to the labelling for Humira®. If the result is positive, patients may participate in the trial if further work up (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active TB. If latent TB is confirmed, then treatment must have been initiated before treatment in the study and continued according to local country guidelines.
* Known clinically significant (per Investigator opinion) coronary artery disease, significant cardiac arrhythmias, moderate to severe congestive heart failure (New York Heart Association Classes III or IV) or interstitial lung disease observed on chest X-ray.
* Patients with a history of any clinically significant adverse reaction (including serious allergic reactions, or anaphylactic reaction, or hypersensitivity) to murine or chimeric proteins, previously used biological drug or its excipients, or natural rubber and latex.
* Positive serology for HBV or HCV.
* Receipt of a live/attenuated vaccine within 12 weeks prior to the Screening Visit; patients who are expecting to receive any live/attenuated virus or bacterial vaccinations during the trial or up to 3 months after the last dose of trial drug.
* Any treatment (including biologic therapies) that, in the opinion of the Investigator, may place the patient at unacceptable risk during the trial.
* Known active infection of any kind (excluding fungal infections of nail beds), any major episode of infection requiring hospitalisation or treatment with intravenous (i.v.) antiinfectives within 4 weeks of the Screening Visit or completion of oral anti-infectives within 2 weeks of the Screening Visit.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 times upper limit of normal (ULN) at screening.
* Hemoglobin < 8.0 g/dL at screening.
* Platelets < 100,000/μL at screening.
* Leukocyte count < 4000/μL at screening.
* Calculated creatinine clearance < 60 mL/min at screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (21):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Dermatology Research Associates, Los Angeles, California
  - Shahram Jacobs MD, Inc./Unison Clinical Trials, Sherman Oaks, California
  - Universal Clinical Research, Hialeah, Florida
  - New Horizon Research Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Progressive Medical Research, Port Orange, Florida
  - University of South Florida, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Dermatology Consulting Services, High Point, North Carolina
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Palmetto Clinical Trial Services, LLC, Fountain Inn, South Carolina
  - Arlington Research Center, Arlington, Texas
  - Center for Clinical Studies, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
- Germany (2):
  - Rothhaar Studien GmbH, Berlin
  - Klinische Forschung Dresden, GmbH, Dresden
- Hungary (3):
  - UNO Medical Trials Kft., Budapest
  - Szabolcs-Szatmar-Bereg Univ.teach.Hosp, Nyíregyháza
  - ALLERGO-DERM BAKOS Kft., Szolnok
- Latvia (6):
  - Riga 1st Hosp, Out-patient Department, Riga
  - Derma Clinic Riga Ltd, Riga
  - Health Center 4, Affiliate Diagnostic Center, Riga
  - J. Kisis Ltd, Riga
  - Smite Aija practice in dermatology and venerology, Talsi
  - Outpatient Clinic of Ventspils, Ventspils
- Poland (10):
  - Poradnia Kardiologiczna Jaroslaw Jurowiecki, Gdansk
  - Synexus Polska SCM Sp. z o.o. Gdansku, Gdansk, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia, Gdynia
  - Malopolskie medical center S.C, Krakow, Krakow
  - SANTA FAMILIA Centrum Badan, Profilaktyki i Leczenia, Lodz
  - Dermoklinika medical center, Lodz, Lodz
  - Medicome Sp. z o.o., Oświęcim
  - Clinmedica Research Omc sp. z o.o. sp.k., Skierniewice, Skierniewice
  - Laser Clin. S.C. Dr T. Kochanowski Dr A. Krolicki, Szczecin, Szczecin
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warszawa, Warsaw
- Russia (3):
  - LLC "Alliance Biomedical - Russian Group", Saint Petersburg
  - EKO-Bezopasnost, St. Petersburg, Saint Petersburg
  - Institution of Healthcare "Nikolaevskaya Hospital", Saint Petersburg
- Ukraine (4):
  - SI Road Clinical Hospital of DS of SE PZ Dept of Dermatovenerology SI DMA of MOHU, Dnipro
  - Kherson clin.hosp.Afanasiia&Olhy Tropinykh, Kherson
  - Treatment - Diagnostic Center PE Asclepius, Uzhhorod
  - CI Zaporizhzhia Regional Dermatovenerologic Clinical Dispensary of Zaporizhzhia RC, Zaporizhzhia

REFERENCES:
- [Derived] Menter A, Cohen S, Kay J, Strand V, Gottlieb A, Hanauer S, Eduru SK, Buschke S, Lang B, Liesenfeld KH, Schaible J, McCabe D. Switching Between Adalimumab Reference Product and BI 695501 in Patients with Chronic Plaque Psoriasis (VOLTAIRE-X): A Randomized Controlled Trial. Am J Clin Dermatol. 2022 Sep;23(5):719-728. doi: 10.1007/s40257-022-00708-w. Epub 2022 Aug 7. PMID 35934770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 58-week, multiple-dose, active comparator trial of BI 695501 and US-licensed Humira in patients with moderate to severe chronic plaque psoriasis. The trial consisted of a single-arm run-in period of 14 weeks for all patients, followed by a randomized, double-blind, 2-arm period of 34 weeks. The total treatment period was 48 weeks followed by 10 weeks of safety follow up (SFU).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Not Randomized: Patients received US-licensed Humira during the run-in period. A loading dose of 80 milligrams (mg) US-licensed Humira on Day 1 (Week 1), followed by 40 mg every other week from Week 2 to Week 12. At the beginning of Week 14, patients who achieved at least a 50 percent reduction in Psoriasis Area and Severity Index (PASI50) response were randomized in a 1:1 ratio to either a continuous arm receiving 40mg of US-licensed Humira every other week until week 48 or in a switching arm separated in 3 periods.
  Patients who participated in the run-in period but not being randomized after run-in period were included in this group.
- Switching Arm (Post-Randomization Period): Patients initially received US-licensed Humira during the run-in period (Period 1) of 14 weeks and were then randomized to the switching arm for the randomized treatment period (Period 2) of 34 weeks followed by 10 weeks of safety follow-up.
  During Period 1, patients were administered with a loading dose of 80 milligram (mg) US-licensed Humira on Day 1 (Week 1), followed by 40 mg every other week from Week 2 to Week 12. During Period 2, patients received 40 mg BI 695501 at Week 14 and Week 16 (2 injections), followed by 40 mg US-licensed Humira at Week 18 and Week 20 (2 injections), and subsequently 40 mg BI 695501 every other week from Week 22 to Week 48 (14 injections). Trial medication were administered by subcutaneous (s.c.) injection providing in single-use pre-filled syringes (PFS) containing 40 mg of adalimumab or BI 695501 per 0.8 milliliter (mL).
  Patients who went through the run-in period and being randomised into the switching arm were included in this group.
- Continuous Humira (Post-Randomization Period): Patients initially received US-licensed Humira during the run-in period of 14 weeks (Period 1) and were then randomized to the continuous Humira arm for the randomized treatment period of 34 weeks (Period 2) followed by 10 weeks of safety follow-up. During Period 1, patients were administered with a loading dose of 80 milligram (mg) US-licensed Humira on Day 1 (Week 1), followed by 40 mg every other week from Week 2 to Week 12. During Period 2, patients received 40 mg US-licensed Humira every other week from Week 14 to Week 48 (18 injections).Trial medication were administered by subcutaneous (s.c.) injection providing in single-use pre-filled syringes (PFS) containing 40 mg of adalimumab per 0.8 milliliter (mL).
  Patients who went through the run-in period and being randomised into the continuous Humira arm were included in this group.
Period: 12-Week Run-in Period
Arm/Group | Not Randomized | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
Started (Enrolled) | 21 | 118 | 120
Completed (Completed the run-in period) | 0 | 118 | 120
Not Completed | 21 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Lack of Efficacy | 6 | 0 | 0
Period: 48-Week Randomized Responder Period
Arm/Group | Not Randomized | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
Started (Randomization) | 0 | 118 | 120
Completed (Completed the trial) | 0 | 107 | 91
Not Completed | 0 | 11 | 29
Not completed — Missed study visit | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 3 | 8
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 5 | 17
Not completed — Adverse Event | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) contained all randomized patients who received at least 1 dose of trial medication administered in the post-randomization period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period) | Total
Number analyzed (Participants) | 118 | 120 | 238
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.1 (13.95) | 43.7 (13.69) | 44.9 (13.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 44 | 81
  Male | 81 | 76 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 18 | 36
  Not Hispanic or Latino | 100 | 102 | 202
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 0 | 2
  White | 113 | 119 | 232
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time Curve Over the Dosing Interval of Week 30 to 32 (AUCτ, 30-32) for Adalimumab in Plasma
Description: Area Under the Plasma Concentration Time Curve Over the 2 weeks dosing Interval between Week 30 to 32 (AUCτ, 30-32) for Adalimumab in plasma was reported.
Time Frame: Pre-dose at Week 30, at 72, 120, 168 and 240 hours after the Week 30 dosing, and pre-dose at Week 32.
Population: The Pharmacokinetic (PK) Set (PKS) included all patients from the TS who provided at least 1 primary PK parameter that was not excluded due to a protocol violation relevant to the evaluation of PK.
Measure: Mean (Standard Deviation); unit: microgram * hours / milliliter
Arm/Group | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
Number analyzed (Participants) | 102 | 93
microgram * hours / milliliter | 2040 (1420) | 1980 (1600)
Statistical Analysis 1: Comparison: Switching Arm (Post-Randomization Period) vs Continuous Humira (Post-Randomization Period); The null hypothesis was that the ratio of expected means for Switching vs. Continuous Humira is less than 80.00% or more than 125.00%; Test type: Equivalence — Equivalence was concluded if the confidence interval (CI) for the least squares (LS) means ratio was included in the pre-defined equivalence range of 80.00% to 125.00%; Least squares means ratio = 105.19, 90.2% CI 2-sided [96.58 to 114.64] — The least squares means were from ANCOVA. Ratio was calculated with the switching arm in the numerator and the continuous arm in the denominator

2. Primary Outcome: Maximum Observed Concentration During the Dosing Interval Week 30-32 (Cmax, 30-32) for Adalimumab in Plasma
Description: Maximum observed concentration during the 2 weeks dosing interval between Week 30 to 32 (Cmax, 30-32) for Adalimumab in plasma was reported.
Time Frame: Pre-dose at Week 30, at 72, 120, 168 and 240 hours after the Week 30 dosing, and pre-dose at Week 32.
Population: The PK Set (PKS) included all patients from the TS who provided at least 1 primary PK parameter that was not excluded due to a protocol violation relevant to the evaluation of PK.
Measure: Mean (Standard Deviation); unit: microgram / milliliter
Arm/Group | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
Number analyzed (Participants) | 104 | 99
microgram / milliliter | 7.13 (4.63) | 7.14 (5.37)
Statistical Analysis 1: Comparison: Switching Arm (Post-Randomization Period) vs Continuous Humira (Post-Randomization Period); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Equivalence was concluded if the confidence interval (CI) for the LS means ratio was included in the pre-defined equivalence range of 80.00% to 125.00%; Least squares means ratio = 101.14, 90.2% CI 2-sided [93.26 to 109.70] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Minimum Observed Concentration During the Dosing Interval of Week 30 to 32 (Cmin, 30-32) for Adalimumab in Plasma
Description: Minimum Observed Concentration During the 2 weeks Dosing Interval between Week 30 to 32 (Cmin, 30-32) for Adalimumab in plasma was reported.
Time Frame: Pre-dose at Week 30, at 72, 120, 168 and 240 hours after the Week 30 dosing, and pre-dose at Week 32.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micogram / milliliter
Arm/Group | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
Number analyzed (Participants) | 104 | 98
micogram / milliliter | 5.04 (3.89) | 4.66 (4.19)
Statistical Analysis 1: Comparison: Switching Arm (Post-Randomization Period) vs Continuous Humira (Post-Randomization Period); No hypothesis was defined and no statistical test was performed; Test type: Other; Least squares means ratio = 107.31, 90.2% CI 2-sided [97.33 to 118.43] — The least squares means were from ANCOVA. Ratio was calculated with the switching arm as numerator and the continuous arm as the denominator

4. Secondary Outcome: Time to Maximum Observed Concentration During the Dosing Interval of Week 30 to 32 (Tmax, 30-32) for Adalimumab in Plasma
Description: Time to Maximum Observed Concentration During the 2 weeks Dosing Interval between Week 30 to 32 (tmax, 30-32) for Adalimumab in plasma was reported.
Time Frame: Pre-dose at Week 30, at 72, 120, 168 and 240 hours after the Week 30 dosing, and pre-dose at Week 32.
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
Number analyzed (Participants) | 104 | 99
hours | 72.7 [66.0 to 336] | 72.3 [46.8 to 240]

5. Secondary Outcome: Percentage of Patients With a 75% Reduction in Psoriasis Area and Severity Index (PASI75) Response at Week 32
Description: The PASI is an established measure of clinical efficacy for psoriasis medications. The PASI is a tool which provides a numeric scoring for patients' overall psoriasis disease state, with scores ranging from 0 to 72. It is a linear combination of percent of surface area of skin that is affected and the severity of erythema, induration, and desquamation over four body regions (head, trunk, upper extremities and lower extremities). Higher PASI scores indicate more severe psoriasis. PASI is generally summarized as a dichotomous outcome based on achieving over an X percent(%) reduction from baseline (or PASIX), where X is 50, 75, 90, and 100. Results are reported for percentage of patients with a PASI75 response at Week 32. Analysis was done on per-protocol analysis set (PPS).
Time Frame: At week 32
Population: The PPS contained all patients from the TS who did not experience any important protocol violations relevant for efficacy. Missing data were imputed via non-responder imputation for patients who discontinued treatment early and multiple imputation (MI) for missing at random value. There were no cases where it was required to implement MI.
Measure: Number; unit: Percentage of patients
Arm/Group | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
Number analyzed (Participants) | 118 | 119
Percentage of patients | 84.75 | 78.99
Statistical Analysis 1: Comparison: Switching Arm (Post-Randomization Period) vs Continuous Humira (Post-Randomization Period); No hypothesis was tested; Test type: Other; Risk Difference (RD) = 5.75, 90% CI 2-sided [-2.45 to 13.96] — Risk difference was calculated as Switching arm minus Continuous Humira

6. Secondary Outcome: Percentage of Patients With a Static Physician's Global Assessment (sPGA) Score ≤ 1 (Clear or Almost Clear) at Week 32
Description: The sPGA is a 5-point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. The assessment is considered "static", which refers to the patient's disease state at the time of the assessments, without comparison to any of the patient's previous disease states (dynamic), whether at baseline or at a previous visit. A lower score indicates less body coverage and a higher score indicates more severe disease (0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe). Results are reported for percentage of patients with a sPGA score of ≤ 1 (clear or almost clear) at Week 32. Analysis was done on per-protocol analysis set (PPS).
Time Frame: At week 32
Population: as for outcome 5
Measure: Number; unit: Percentage of patients
Arm/Group | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
Number analyzed (Participants) | 118 | 119
Percentage of patients | 70.34 | 64.71
Statistical Analysis 1: Comparison: Switching Arm (Post-Randomization Period) vs Continuous Humira (Post-Randomization Period); No hypothesis was tested; Test type: Other; Risk Difference (RD) = 5.63, 90% CI 2-sided [-4.35 to 15.62] — Risk difference was calculated as Switching arm minus Continuous Humira

7. Secondary Outcome: Number of Patients With Anti-drug Antibody (ADA) to Adalimumab at Week 32
Description: Number of patients with a confirmed positive anti-drug antibody (ADA) response to Adalimumab (BI 695501 or Humira) at Week 32. A participant was considered "ADA positive" if the blank normalized signal in the ADA screening assay was equal to or above the study specific ADA screening cut point factor of 1.06 and the signal inhibition by drug in the ADA confirmatory assay was equal to or above the study specific ADA confirmatory cut points (11.4% for signal inhibition with Humira and 12.0% for signal inhibition with BI 695501).
Time Frame: Immunogenicity samples were collected pre-dose at Week 32.
Population: Patients in the TS who had non-missing endpoints. The TS contained all randomized patients who received at least 1 dose of trial medication administered in the post-randomization period.
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
Number analyzed (Participants) | 112 | 112
Participants
  Negative | 11 | 6
  Positive | 101 | 104
  Total reportable | 112 | 110
  Not reportable | 0 | 2

8. Secondary Outcome: Number of Patients With Neutralizing Antibody (nAb) to Adalimumab at Week 32
Description: Number of patients with a positive neutralizing anti-drug antibody (nAb) response to Adalimumab (BI 695501 or Humira) at Week 32. A participant was considered "nAb positive" if the blank normalized signal in the nAb screening assay was equal to or below the study specific nAb screening cut point factor of 0.836.
Time Frame: Immunogenicity samples were collected pre-dose at Week 32.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
Number analyzed (Participants) | 112 | 112
Participants
  Negative | 66 | 64
  Positive | 46 | 46
  Total reportable | 112 | 110
  Not reportable | 0 | 2

9. Secondary Outcome: Anti-drug Antibody (ADA) Titer of Patients With ADA at Week 32
Description: Anti-drug antibody (ADA) titer of patients with a confirmed positive ADA response to Adalimumab (BI 695501 or Humira) at Week 32.
Time Frame: Immunogenicity samples were collected pre-dose at Week 32.
Population: Analysis was on patients in the treated set (TS) with positive ADA at week 32. The TS contained all randomized patients who received at least 1 dose of trial medication administered in the post-randomization period.
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
Number analyzed (Participants) | 101 | 104
Titer | 64.0 [32.00 to 256.00] | 128 [16.00 to 256.00]

10. Secondary Outcome: Neutralizing Anti-drug Antibody (nAb) Titer of Patients With nAb at Week 32
Description: Neutralizing anti-drug antibody (nAb) titer of patients with a positive nAb response to Adalimumab (BI 695501 or Humira) at Week 32.
Time Frame: Immunogenicity samples were collected pre-dose at Week 32.
Population: Analysis was on patients in the treated set (TS) with positive nAb at week 32. The TS contained all randomized patients who received at least 1 dose of trial medication administered in the post-randomization period.
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
Number analyzed (Participants) | 46 | 46
Titer | 2.0 [1.00 to 4.00] | 2.0 [1.00 to 2.00]

11. Secondary Outcome: Percentage of Patients With Drug-related Adverse Events (AEs) During the Post-Randomization Period
Description: Analysis of AEs focused on treatment-emergent adverse events (TEAEs) and is presented here for the post-randomization period (Week 14 to 58). For the post-randomization period analysis, TEAEs were defined as AEs that started or worsened on or after the first dose of trial post-randomization medication and prior to the last dose of trial post-randomization medication + 10 weeks.
Time Frame: From first dose of trial post-randomization medication until 10 weeks after last dose of trial post-randomization medication, up to 44 weeks
Population: The Treated Set (TS) contained all randomized patients who received at least 1 dose of trial medication administered in the post-randomization period.
Measure: Number; unit: Percentage of patients
Arm/Group | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
Number analyzed (Participants) | 118 | 120
Percentage of patients | 11.9 | 18.3

ADVERSE EVENTS:
Time Frame: From first post-randomized trial medication until 10 weeks after last dose, up to 44 weeks (Post-Randomization Period). From first dose of Humira and prior to the first dose of post-randomization medication+10 weeks, up to 24 weeks (Run-In Period).
Description: Safety analyses were performed based on the Treated Set (TS) and Run-in Treated Set (RTS). The TS contained all randomized patients who received at least 1 dose of trial medication administered in the post-randomization period. The RTS contained all enrolled patients treated with at least 1 dose of US-licensed Humira during the run-in period.
Groups:
- Humira Containing All RTS Subjects (Run-In Period): All patients received US-licensed Humira during the run-in period of 14 weeks (Period 1). Patients were administered with a loading dose of 80 milligram (mg) US-licensed Humira on Day 1 (Week 1), followed by 40 mg every other week from Week 2 to Week 12. Trial medication were administered by subcutaneous (s.c.) injection providing in single-use pre-filled syringes (PFS) containing 40 mg of adalimumab per 0.8 milliliter (mL).
  All patients in the run-in period were in this group including those who were randomised and who did not being randomised after the run-in period.
Arm/Group | Humira Containing All RTS Subjects (Run-In Period) | Switching Arm (Post-Randomization Period) | Continuous Humira (Post-Randomization Period)
All-Cause Mortality (participants affected / at risk) | 1/259 | 0/118 | 0/120
Serious Adverse Events (participants affected / at risk) | 6/259 | 5/118 | 4/120
Other Adverse Events (participants affected / at risk) | 24/259 | 17/118 | 11/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Humira Containing All RTS Subjects (Run-In Period) (N=259) | Switching Arm (Post-Randomization Period) (N=118) | Continuous Humira (Post-Randomization Period) (N=120)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Sinus arrest (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Pneumonia chlamydial (Infections and infestations) | 0 | 0 | 1
Diffuse axonal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Demyelination (Nervous system disorders) | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Humira Containing All RTS Subjects (Run-In Period) (N=259) | Switching Arm (Post-Randomization Period) (N=118) | Continuous Humira (Post-Randomization Period) (N=120)
Nasopharyngitis (Infections and infestations) | 16 | 11 | 5
Headache (Nervous system disorders) | 10 | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT03210259/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT03210259/SAP_001.pdf